CLINICAL TRIAL: NCT07138079
Title: The Comparison of the Effectiveness of the Self-Pressurizing Air-Q Intubating Laryngeal Airway in Totally Edentulous and Dentate Geriatric Patients
Brief Title: Air-Q in Totally Edentulous and Dentate Geriatric Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeynep Koc, principal investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ZeynepKoc004
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Complications; Sore-throat
Keywords: Air-Q Laryngeal İntubating Airway; Oropharyngeal leak pressure; supraglottic airways; Edentulous patients; Geriatric patients
MeSH Terms: conditions — Postoperative Complications; Pharyngitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- edentulous group (Active Comparator): under general anesthesia, edentulous geriatric patients inserted Air- Q intubating airway
  Interventions: Other: edentulous geriatric patients
- gentate group (Active Comparator): under general anesthesia, dantate geriatric patients inserted Air- Q intubating airway
  Interventions: Other: dentate geriatric patients

INTERVENTIONS:
Other: edentulous geriatric patients — Edentulous geriatric patients will be inserted Air-Q Intubating Airway under general anesthesia.
  Arms: edentulous group
Other: dentate geriatric patients — Dentate geriatric patients will be inserted Air-Q Intubating Airway under general anesthesia.
  Arms: gentate group

SUMMARY:
In this study, we aim to investigate the clinical performance, efficacy, and associated complications of the Air-Q Intubating Laryngeal Airway in totally edentulous and dentate geriatric patients.

DETAILED DESCRIPTION:
In the elderly population, the prevalence of totally edentulous patients over the age of 65 exceeds 60%. With aging, parapharyngeal fat deposition increases and contributes to pharyngeal collapse in elderly patients . In elderly patients with total tooth loss, face mask ventilation is difficult because standard face masks do not fit well on edentulous faces. Additionally, during general anesthesia, loss of muscle tone, reduced oropharyngeal air space, posterior displacement of the tongue, and airway obstruction caused by the soft palate and epiglottis all make ventilation challenging . Structural changes in the airway, combined with age-related physiological alterations in respiration, may reduce oxygen saturation, blunt the hypoxic response, and increase the risk of postoperative respiratory complications. Due to age-related acquired changes in pharyngeal muscle activity, the likelihood of skeletal structural abnormalities such as retrognathia-often associated with difficult airways-has been proposed (2). Therefore, these age-related changes may influence the clinical performance of supraglottic airway devices (SADs).

Recently, SADs that do not require manual cuff inflation have gained popularity in various clinical settings due to their advantage of eliminating the need for manual cuff inflation and cuff pressure monitoring (5,6). The Air-Q is a supraglottic airway device that connects to an airway tube through a communication port, allowing self-pressurization of the cuff in response to airway pressure.

In this study, we aim to investigate the clinical performance, efficacy, and associated complications of the Air-Q Intubating Laryngeal Airway in totally edentulous and dentate geriatric patients.

ELIGIBILITY:
Inclusion Criteria:

* 65-90 year-old patients
* Edentulous and gentate patients
* American Society of Anesthesiologist Physical Status classification I-III,
* Undergoing an elective operation under general anesthesia in our hospital

Exclusion Criteria:

* Predicted difficult airway (Mallampati class 4, mouth opening < 3 cm, or thyromental distance < 6 cm)
* Body mass index (BMI) > 40 kg/m2
* Patients with a high risk of aspiration (e.g., history of gastrectomy, -gastroesophageal reflux disease, or hiatal hernia),
* Unstable vital signs
* Cervical spine problems, Respiratory complications (e.g. recent pneumonia).

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2025-09-29 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of oropharyngeal leak pressure (OLP) | One minute after successful LMA placement
  One minute after successful LMA placement and fixation, oropharyngeal leak pressure

SECONDARY OUTCOMES:
Air-Q insertion time | 3 minutes after induction of anesthesia
  Successful Air-Q placement will be confirmed by visualizing a square waveform on the ventilator and observing chest wall movement.
ease of SGA placement | 3 minutes after induction of anesthesia
  Successful SGA placement will be confirmed by visualizing a square waveform on the ventilator and observing chest wall movement.
maneuvers required for successful ventilation | 3 minutes after induction of anesthesia
  It will be recorded whether any further maneuvers are required: Gentle pushing or pulling of the LMA to adjust its depth, jaw-thrust maneuver, and flexion or extension of the head.
fiberoptic view grading | 3 minutes after induction of anesthesia
  The Brimacombe score will be used to evaluate the view obtained with fiberoptic bronchoscopy. 1: Vocal cords are not visible; 2: Vocal cords and anterior epiglottis are visible; 3: Vocal cords and posterior epiglottis are visible; 4: Vocal cords are visible.

OTHER OUTCOMES:
Complications during Air-Q removal (emerge) | One minute after Air-Q removal
  Complications during SP_Air-Q and proseal LMA removal (emerge) such as breath-holding during emergence, airway obstruction, coughing, hypoxia (SpO2 < 90%), vomiting, lip-tongue-teeth trauma, and bleeding, will be recorded.
Sore throat | 1 hour postoperatively
  The presence or absence of sore throat will be recorded at the 24th postoperative hour
Sore throat | 24 hours postoperatively
  The presence or absence of sore throat will be recorded at the 24th postoperative hour
dysphonia | 1 hour postoperatively
  The presence or absence of dysphonia will be recorded at the firsth postoperative hour
dysphonia | 24 hours postoperatively
  The presence or absence of dysphonia will be recorded at the firsth postoperative hour

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Koç, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beydes T, Kucukguclu S, Ozbilgin S, Kuvaki B, Ademoglu M, Sari M. Comparison of Laryngeal Mask Airway Supreme(TM) Versus Unique(TM) in Edentulous Geriatric Patients. Turk J Anaesthesiol Reanim. 2016 Feb;44(1):32-6. doi: 10.5152/TJAR.2016.22129. Epub 2016 Feb 1. PMID 27366552
- [Background] Genez M, Kucukguclu S, Ozbilgin S, Kuvaki B, Beydes T, Aksoy Sari M. A comparison of usage of the laryngeal mask UniqueTM in denticulate and edentulate geriatric patients. Turk J Med Sci. 2017 Jun 12;47(3):854-860. doi: 10.3906/sag-1603-206. PMID 28618734
- [Background] Lee JS, Kim DH, Choi SH, Ha SH, Kim S, Kim MS. Prospective, Randomized Comparison of the i-gel and the Self-Pressurized air-Q Intubating Laryngeal Airway in Elderly Anesthetized Patients. Anesth Analg. 2020 Feb;130(2):480-487. doi: 10.1213/ANE.0000000000003849. PMID 30320644